CLINICAL TRIAL: NCT04277871
Title: Effects of an Intervention on Improving Midlife Women's Menopause-related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-2314-B-038-039
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Genitourinary Symptoms
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group received an educational section and related educational materials. The educational section involved two sub-sections: a discussion section and an abbreviated practice section. The intervention group attended on-site group practice sections and performed individual home-based practice.
  Interventions: Behavioral: Pelvic floor muscles training (PFMT) combined with yoga
- The comparison group (Active Comparator): The comparison group received an educational section and related educational materials. The educational section involved two sub-sections: a discussion section and an abbreviated practice section. The comparison group performed individual home-based practice only.
  Interventions: Behavioral: Pelvic floor muscles training (PFMT) combined with yoga

INTERVENTIONS:
Behavioral: Pelvic floor muscles training (PFMT) combined with yoga — All study participants were instructed to perform PFMT combined with yoga with an expectation of performing a 70-minute practice section 3 days in a week. All study participants received a booklet with menopause-related information, a booklet plus an instructional Digital Video Disc for PFMT and yoga practice.

SUMMARY:
This study was an experimental study with repeated measures. Study aims were to examine the effects of pelvic floor muscles training (PFMT) combined with yoga on improving genitourinary/climacteric symptoms, the pelvic floor muscles strength, and health-related quality of life (HRQL). Study participants were assigned to the intervention group or comparison group. Data analyses were based on the information obtained from 91 midlife women with a mean age of 56.6 years. Information related o the pelvic floor muscles strength was only obtained from 45 women. Descriptive statistics were used to represent study participants' individual characteristics, genitourinary/climacteric symptoms, the pelvic floor muscles strength, and HRQL. Paired t tests, independent t tests, and Generalized Estimating Equation (GEE) procedures were used to examine the intervention effects.

DETAILED DESCRIPTION:
This study was an experimental study with repeated measures. Study aims were to examine the effects of PFMT combined with yoga on improving genitourinary/climacteric symptoms, the pelvic floor muscles strength, and HRQL. Study participants were randomly assigned to the intervention group or comparison group. All study participants received an educational section (a discussion section and an abbreviated practice section) and related educational materials. The intervention group attended on-site group practice sessions and performed individual home-based practice. The comparison group performed individual home-based practice only. Data analyses were based on the information obtained from a sample of midlife women with a mean age of 56.6 years. Relevant information was mainly collected by a structured questionnaire. Information related to the pelvic floor muscles strength was only obtained from 45 women in the intervention group by using the FemiScan pelvic floor therapy system. Descriptive statistics were used to represent study participants' individual characteristics, genitourinary/climacteric symptoms, the pelvic floor muscles strength, and HRQL. Paired t tests, independent t tests, and GEE procedures were used to examine the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Women who experienced ≥1 genitourinary symptoms.

Exclusion Criteria:

* Being pregnancy or breastfeeding, experiencing iatrogenic menopause (e.g., surgery, chemotherapy or radiation related), maintaining regular PFMT and/or yoga practices, using oral contraceptive or psychiatric medications, and having physical weakness/limitation or major cognitive impairment.

Ages: 47 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Genitourinary Symptoms | Baseline
  Self-reporting 11 genitourinary symptoms: We generated three items to measure genital symptoms based on available information (The North American Menopause Society, 2013), and used the Lower Urinary Tract Symptoms (LUTS) subscale in the Taiwan Teacher Bladder Survey for measuring LUTS (Liao et al., 2006).
Genitourinary Symptoms | 3-month follow-up
  Self-reporting 11 genitourinary symptoms: We generated three items to measure genital symptoms based on available information (The North American Menopause Society, 2013), and used the Lower Urinary Tract Symptoms (LUTS) subscale in the Taiwan Teacher Bladder Survey for measuring LUTS (Liao et al., 2006).
Genitourinary Symptoms | 6-month follow-up
  Self-reporting 11 genitourinary symptoms: We generated three items to measure genital symptoms based on available information (The North American Menopause Society, 2013), and used the Lower Urinary Tract Symptoms (LUTS) subscale in the Taiwan Teacher Bladder Survey for measuring LUTS (Liao et al., 2006).
Genitourinary Symptoms | 9-month follow-up
  Self-reporting 11 genitourinary symptoms: We generated three items to measure genital symptoms based on available information (The North American Menopause Society, 2013), and used the Lower Urinary Tract Symptoms (LUTS) subscale in the Taiwan Teacher Bladder Survey for measuring LUTS (Liao et al., 2006).
Genitourinary Symptoms | 12-month follow-up
  Self-reporting 11 genitourinary symptoms: We generated three items to measure genital symptoms based on available information (The North American Menopause Society, 2013), and used the Lower Urinary Tract Symptoms (LUTS) subscale in the Taiwan Teacher Bladder Survey for measuring LUTS (Liao et al., 2006).
Climacteric Symptoms | Baseline
  Self-reporting 21 physical and psychological symptoms: We used the Taiwan-version of the Greene Climacteric Scale for measuring climacteric symptoms (Greene, 2008).
Climacteric Symptoms | 3-month follow-up
  Self-reporting 21 physical and psychological symptoms: We used the Taiwan-version of the Greene Climacteric Scale for measuring climacteric symptoms (Greene, 2008).
Climacteric Symptoms | 6-month follow-up
  Self-reporting 21 physical and psychological symptoms: We used the Taiwan-version of the Greene Climacteric Scale for measuring climacteric symptoms (Greene, 2008).
Climacteric Symptoms | 9-month follow-up
  Self-reporting 21 physical and psychological symptoms: We used the Taiwan-version of the Greene Climacteric Scale for measuring climacteric symptoms (Greene, 2008).
Climacteric Symptoms | 12-month follow-up
  Self-reporting 21 physical and psychological symptoms: We used the Taiwan-version of the Greene Climacteric Scale for measuring climacteric symptoms (Greene, 2008).

SECONDARY OUTCOMES:
The Pelvic Floor Muscles Strength | Baseline
  For the intervention group, we obtained the Pelvic Floor Muscles' perianal surface electromyography by using the FemiScan pelvic floor therapy system. Two parameters (activity and peak; µV) resulted from the electromyography were used to represent the Pelvic Floor Muscles strength (Mega Electronics Ltd, 2002-2006).
The Pelvic Floor Muscles Strength | 3-month follow-up
  For the intervention group, we obtained the Pelvic Floor Muscles' perianal surface electromyography by using the FemiScan pelvic floor therapy system. Two parameters (activity and peak; µV) resulted from the electromyography were used to represent the Pelvic Floor Muscles strength (Mega Electronics Ltd, 2002-2006) .
The Pelvic Floor Muscles Strength | 6-month follow-up
  For the intervention group, we obtained the Pelvic Floor Muscles' perianal surface electromyography by using the FemiScan pelvic floor therapy system. Two parameters (activity and peak; µV) resulted from the electromyography were used to represent the Pelvic Floor Muscles strength (Mega Electronics Ltd, 2002-2006).
The Pelvic Floor Muscles Strength | 9-month follow-up
  For the intervention group, we obtained the Pelvic Floor Muscles' perianal surface electromyography by using the FemiScan pelvic floor therapy system. Two parameters (activity and peak; µV) resulted from the electromyography were used to represent the Pelvic Floor Muscles strength (Mega Electronics Ltd, 2002-2006).
The Pelvic Floor Muscles Strength | 12-month follow-up
  For the intervention group, we obtained the Pelvic Floor Muscles' perianal surface electromyography by using the FemiScan pelvic floor therapy system. Two parameters (activity and peak; µV) resulted from the electromyography were used to represent the Pelvic Floor Muscles strength (Mega Electronics Ltd, 2002-2006).

OTHER OUTCOMES:
Health-related Quality of Life | Baseline
  We used the Taiwan version of the Short Form-36 (SF-36) Health Survey to measure quality of life (Fuh et al., 2000).
Health-related Quality of Life | 3-month follow-up
  We used the Taiwan version of the Short Form-36 (SF-36) Health Survey to measure quality of life (Fuh et al., 2000).
Health-related Quality of Life | 6-month follow-up
  We used the Taiwan version of the Short Form-36 (SF-36) Health Survey to measure quality of life (Fuh et al., 2000).
Health-related Quality of Life | 9-month follow-up
  We used the Taiwan version of the Short Form-36 (SF-36) Health Survey to measure quality of life (Fuh et al., 2000).
Health-related Quality of Life | 12-month follow-up
  We used the Taiwan version of the Short Form-36 (SF-36) Health Survey to measure quality of life (Fuh et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Mei Liao, PhD, Principal Investigator — National Yang-Ming University, Taiwan, R.O.C

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Cramer H, Peng W, Lauche R. Yoga for menopausal symptoms-A systematic review and meta-analysis. Maturitas. 2018 Mar;109:13-25. doi: 10.1016/j.maturitas.2017.12.005. Epub 2017 Dec 6. PMID 29452777
- [Background] Sha K, Palmer MH, Yeo S. Yoga's Biophysiological Effects on Lower Urinary Tract Symptoms: A Scoping Review. J Altern Complement Med. 2019 Mar;25(3):279-287. doi: 10.1089/acm.2018.0382. Epub 2019 Feb 8. PMID 30735055
- [Background] Mercier J, Morin M, Zaki D, Reichetzer B, Lemieux MC, Khalife S, Dumoulin C. Pelvic floor muscle training as a treatment for genitourinary syndrome of menopause: A single-arm feasibility study. Maturitas. 2019 Jul;125:57-62. doi: 10.1016/j.maturitas.2019.03.002. Epub 2019 Mar 29. PMID 31133219
- [Background] Kim GS, Kim EG, Shin KY, Choo HJ, Kim MJ. Combined pelvic muscle exercise and yoga program for urinary incontinence in middle-aged women. Jpn J Nurs Sci. 2015 Oct;12(4):330-9. doi: 10.1111/jjns.12072. Epub 2015 Feb 23. PMID 25705816
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 2008 Sep-Oct;61(1-2):78-84. doi: 10.1016/j.maturitas.2008.09.011. PMID 19434881
- [Background] Liao YM, Dougherty MC, Boyington AR, Lynn MR, Palmer MH. Developing and validating a Chinese instrument to measure lower urinary tract symptoms among employed women in Taiwan. Nurs Outlook. 2006 Nov-Dec;54(6):353-61. doi: 10.1016/j.outlook.2006.09.003. PMID 17142154
- [Background] Fuh JL, Wang SJ, Lu SR, Juang KD, Lee SJ. Psychometric evaluation of a Chinese (Taiwanese) version of the SF-36 health survey amongst middle-aged women from a rural community. Qual Life Res. 2000;9(6):675-83. doi: 10.1023/a:1008993821633. PMID 11236857
- [Background] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Am J Obstet Gynecol. 2002 Jul;187(1):116-26. doi: 10.1067/mob.2002.125704. No abstract available. PMID 12114899